CLINICAL TRIAL: NCT02242448
Title: Imaging Techniques in CT: Technical Development
Status: Terminated | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Other Study IDs: 140158; 14-CC-0158
Record Dates: First submitted 2014-07-31; First posted 2014-09-17 (Estimated); Last update posted 2019-12-04 (Actual); Status verified 2019-10-30

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteer; Contrast

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Background:

- Computed tomography (CT) scanning is a procedure that helps doctors with diagnoses. It uses X-ray radiation to produce an image in three dimensions. Researchers want to study how to get the best quality CT scans using the lowest possible radiation dose.

Objective:

- To determine how to improve CT scanning.

Eligibility:

- Adults 45 years of age and older who have not had a CT scan in the past year and do not have kidney disease.

Design:

* Participants will be screened with a medical history and blood and urine tests.
* Nurses will put an intravenous (IV) line into an arm or hand vein. It will stay in for several hours during the magnetic resonance imaging (MRI) and CT scans. Through this IV, blood will be taken, dye will be injected, and medicine will be given.
* Participants may have a CT scan of the heart, head, chest, abdomen, and/or pelvis. Participants will lie on their back on a table. The table will slide into a donut-shaped machine. An X-ray tube will move around the body, taking pictures.
* Participants may be given a drug called a beta blocker by mouth or through the IV tube.
* Participants heart rate and blood pressure will be monitored.
* Participants may have an MRI scan. The MRI is a large hollow tube. The participant will lie on a table that will be moved into the tube, which contains a magnetic field. When the imaging starts, a thumping sound will be heard. Headphones or earplugs will be provided to muffle the sound.
* Participants will give blood samples.

DETAILED DESCRIPTION:
In this protocol, computed tomography (CT) imaging performed on healthy volunteers and subjects with disease will be used to test, develop and optimize CT protocols. The results of this optimization will be used to evaluate the performance of new imaging methods and equipment, and to provide essential ground work for research and development for use in future patient CT studies. CT imaging is a noninvasive technology. As appropriate, MRI scans will be used to compare to CT imaging findings to help validate the CT methods.

ELIGIBILITY:
* INCLUSION CRITERIA:
* For new or healthy volunteers currently participating in an NIH trial: no CT scan in the last year OR For patients enrolled in a treatment or interventional trial at the NIH: no CT scan in the last 6 months
* Lab Eligibility parameters:

  * For CT and MRI contrast enhanced scans:

    ---eGFR greater than or equal to 60 mL/min/1.73m(2) within 7 days prior to scanning
  * For female participants ages 45-60 within 3 days prior to scan (unless post-menopausal or no longer able to bear children, note exemption on initial visit):

    * Pregnancy test result(blood or urine): Negative
* Willing to travel to the NIH for follow-up visits.
* Greater than or equal to 45 years old
* Able to understand and sign informed consent
* Stable clinical status
* Volunteer indicates no history of participation in NIH protocols using research radiation in the last 12 months (e.g. PET research scans, NCI Molecular Imaging Center PET scans, etc)

EXCLUSION CRITERIA:

* Prior CT scan in the last 12 months for new volunteers or healthy volunteers enrolled in NIH trials OR Prior CT scan in the last 6 months for patients enrolled in a treatment or interventional trial
* Pregnant women
* Over 500 lbs and/or a body circumference that prevents the study subject from lying flat in the scanner
* Claustrophobia requiring sedation or anesthesia.
* Known or suspected genetic predisposition to cancer
* Any contraindications that the research team identifies from the subject, radiology department CT and/or MRI questionnaires, and/or History and Assessment.

Exclusion for participation for iodinated contrast for CT

(Inclusive of the above exclusion criteria):

* Allergy to iodinated contrast for scans (study subject will be eligible for non-contrast scans)
* Acute renal failure, renal transplant, dialysis and renal failure (clinically diagnosed).<TAB>
* Lactating women
* Patient preference to not undergo intravenous line placement and/or receive iodinated contrast. Contrast administration is optional and participants may still undergo a non-contrast study.
* Use of metformin-containing products less than 24 hours prior To CT contrast administration
* Other contraindications to iodinated contrast media as determined by the research team.

Exclusion for participation for Gadolinium contrast for MRI

(Inclusive of the above exclusion criteria):

* Allergy to gadolinium for scans using contrast; will be eligible for non-contrast scans.
* Acute renal failure, renal transplant, dialysis and renal failure individuals ( Lab Eligibility parameters and/or clinically diagnosed).<TAB>
* Lactating women
* Patient preference to not undergo intravenous line placement and/or receive gadolinium contrast. Contrast administration is optional and participants may still undergo a non-contrast study.
* Other contraindications to gadolinium contrast media as determined by the research team.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2014-07-31; Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
To enhance imaging quality and safety | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: David A Bluemke, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Halliburton S, Arbab-Zadeh A, Dey D, Einstein AJ, Gentry R, George RT, Gerber T, Mahesh M, Weigold WG. State-of-the-art in CT hardware and scan modes for cardiovascular CT. J Cardiovasc Comput Tomogr. 2012 May-Jun;6(3):154-63. doi: 10.1016/j.jcct.2012.04.005. Epub 2012 Apr 7. PMID 22551595
- [Background] Trattner S, Pearson GDN, Chin C, Cody DD, Gupta R, Hess CP, Kalra MK, Kofler JM Jr, Krishnam MS, Einstein AJ. Standardization and optimization of CT protocols to achieve low dose. J Am Coll Radiol. 2014 Mar;11(3):271-278. doi: 10.1016/j.jacr.2013.10.016. PMID 24589403
- [Background] Mahesh M. Variability in CT protocols. J Am Coll Radiol. 2013 Oct;10(10):805-6. doi: 10.1016/j.jacr.2013.07.005. Epub 2013 Aug 26. No abstract available. PMID 23988585